CLINICAL TRIAL: NCT05694078
Title: Hand Therapy Approach on Lumbrical Muscle Tears in Sport Climbers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hand Therapy Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lumbrical; PhD University Program (Other: Universitat Autonoma de Barcelona)
Record Dates: First submitted 2022-12-23; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Muscle Tear; Hand Injuries; Splints
Keywords: Lumbrical; Sport Climbing; Hand Therapy; Hand Injuries; Relative Motion
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumbrical Injured Climbers (Experimental): 6-weeks relative motion splinting protocol, while pain-free sport activities are permitted
  Interventions: Other: Hand Therapy Splinting Protocol

INTERVENTIONS:
Other: Hand Therapy Splinting Protocol — Relative motion splinting protocol
  Other Names: Relative Motion

SUMMARY:
This study aimes to analyze the effectiveness of a Hand Therapy protocol in the management of patients who suffer from a tear of a lumbrical muscle, regarding on the symptoms during the clinical examination, the disability in their activities of daily living and the sports-specific function.

DETAILED DESCRIPTION:
A prospective intervention study is performed on 50 adult climbers suffering from an injury of the 4th lumbrical muscle. They wear during 3 weeks a 5th finger extension relative motion orthosis, while pain-free sport activities are permitted using a 4th and 5th fingers buddy-taping. After three weeks, patients are told to progressively remove the splint and, after six weeks, the splint is totally removed. Symptoms in the lumbrical stress test are evaluated during the 6 weeks period using dynamometry and goniometry, Finally, Quick-Disabilities of the arm shoulder and hand questionnaire is also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult climbers suffering from an injury of the 4th lumbrical muscle

Exclusion Criteria:

* Patients with previous treatments.
* Patients with concomitant injuries or illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Dinamometry in lumbrical stress test | It will be evaluated at 6 weeks
  Symptoms in the lumbrical stress test will be evaluated during the 6 weeks period using an adapted Jamar handgrip dynamometer on a climbing hold. The climber is told to pull on the hold until the pain starts.

SECONDARY OUTCOMES:
Goniometry in lumbrical stress test | It will be evaluated at 6 weeks
  Finger flexion metacarpophalangeal joint goniometry of the 5th finger is measured during the lumbrical stress test when pain appears
Quick-Disabilities of the arm shoulder and hand questionnaire | It will be evaluated at 6 weeks
  Participants will be asked to answer "Quick-Disabilities of the arm shoulder and hand" questionnaire before the clinical examination. In "Quick-Disabilities of the arm shoulder and hand" each item has response options and, from the item scores, scale scores are calculated, raning from o (no disability) to 100 (most severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Núria Carnicero, Principal Investigator — Hand Therapy Barcelona
Locations (1):
- Hand Therapy Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lutter C, Schweizer A, Schoffl V, Romer F, Bayer T. Lumbrical muscle tear: clinical presentation, imaging findings and outcome. J Hand Surg Eur Vol. 2018 Sep;43(7):767-775. doi: 10.1177/1753193418765716. Epub 2018 Mar 28. PMID 29591320
- [Background] Schweizer A. Lumbrical tears in rock climbers. J Hand Surg Br. 2003 Apr;28(2):187-9. doi: 10.1016/s0266-7681(02)00250-4. PMID 12631495